CLINICAL TRIAL: NCT06897007
Title: Changes in Ciprofol Dosage in Insomnia Patients Undergoing Digestive Endoscopy: a Prospective Cohort Study
Brief Title: Changes in Ciprofol Dosage in Insomnia Patients Undergoing Digestive Endoscopy
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Daxing Teaching Hospital, Capital Medical University (Unknown); Hebei Medical University Third Hospital (Other); Hengshui People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management Affiliation: Beijing Tiantan Hospital, Beijing Tiantan Hospital
Other Study IDs: KY2024-091-02-2
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Insomnia; Digestive Endoscopy
Keywords: Insomnia; Digestive endoscopy; Ciprofol
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Insomnia group: Patients with insomnia
  Interventions: Other: No interventions, it is a observational study
- Normal sleep group: Patients with normal sleep
  Interventions: Other: No interventions, it is a observational study

INTERVENTIONS:
Other: No interventions, it is a observational study — No interventions, this study is to compare the dosage requirement of ciprofol during digestive endoscopy between insomnia group and normal sleep group.

SUMMARY:
To compare the dosage requirement of ciprofol during digestive endoscopy between patients with insomnia and those with normal sleep pattern.

DETAILED DESCRIPTION:
The investigators aim to investigate whether ciprofol dosage requirement is increased in patients with insomnia undergoing digestive endoscopy compared with normal sleep patterns.

ELIGIBILITY:
Inclusion Criteria:

* Patients with insomnia:

  1. Age of 18 - 64 years;
  2. ASA physical status of I - II;
  3. BMI of 15 - 30;
  4. Scheduled for digestive endoscopy under intravenous anesthesia;
  5. Positive screening results according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for insomnia disorder;
  6. 8-item Sleep Condition Indicator (SCI; score 0-4; range 0-32, higher score means better sleep) scored 16 or less;
* Patients with normal sleep:

  1. Age of 18 - 64 years;
  2. ASA physical status of I - II;
  3. BMI of 15 - 30;
  4. Scheduled for digestive endoscopy under intravenous anesthesia;
  5. No history or evidence of insomnia.

Exclusion Criteria:

1. Associated with any neurological disease;
2. Daily alcohol consumption;
3. Any contraindication to intravenous anesthetic drug, such as hypotension or shock;
4. History of allergy to any drug used in the study;
5. Pregnancy or breastfeeding;
6. Patients with sleep apnea syndrome;
7. acute upper respiratory infection;
8. Patients with psychological diseases who report suicidal thoughts;
9. Patients who need to work or take care of children/elderly people frequently at night.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with insomnia and patients with normal sleep patterns
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The total consumption of ciprofol | Up to 1 day
  The total consumption of ciprofol for digestive endoscopy. It includes the total amount of ciprofol required by the patient for the entire process of digestive endoscopy.

SECONDARY OUTCOMES:
The dosage of ciprofol for successful insertion of digestive endoscope | 1 day
  The dosage of ciprofol for successful insertion of digestive endoscope
The occurrence of the respiratory and cardiovascular adverse events | The day for patients undergoing digestive endoscopy and 24 hours after the digestive endoscopy
  The occurrence of the respiratory and cardiovascular adverse events such as hypoxemia, hypotension, hypertension, arrhythmia
The occurrence of the other adverse events | The day for patients undergoing digestive endoscopy and 24 hours after the digestive endoscopy
  The occurrence of the other adverse events such as dizziness, agitation, nausea, vomiting and psychiatric symptom
The incidence of intraoperative recall or awareness | The day for patients undergoing digestive endoscopy and 24 hours after the digestive endoscopy
  The patient is conscious after anesthesia
The recovery time | Up to 1 day
  The time from when the patient stops intravenous anesthetic drug application to when they can open their eyes and nod their heads.
Duration of patients' PACU stay | Up to 1 day
  Patients' stay time in PACU
The ease of operation at this level of sedation evaluated by the gastroenterologists | Up to 1 day
  The ease of operation at this level of sedation (easy/medium/difficult) evaluated by the gastroenterologists
The satisfaction degree of anesthesia effect evaluated by the gastroenterologists | Up to 1 day
  The satisfaction degree of anesthesia effect (satisfactory/medium/unsatisfactory) evaluated by the gastroenterologists
Patients' satisfaction | Up to 1 day
  Patients' satisfaction with the procedure at this level of sedation (satisfactory/medium/unsatisfactory)
Patients' willingness | Up to 1 day
  Patients' willingness to undergo the next procedure at the same level of sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China